CLINICAL TRIAL: NCT02777385
Title: Randomized, Phase II Study Evaluating Concurrent or Sequential Fixed-Dose Pembrolizumab in Combination With Cisplatin and Intensity Modulated Radiotherapy in Intermediate or High Risk, Previously Untreated, Locally Advanced Head and Neck Cancer
Brief Title: Pembrolizumab in Combination With Cisplatin and Intensity Modulated Radiotherapy (IMRT) in Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dan Zandberg (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Dan Zandberg, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 15-132
Record Dates: First submitted 2016-04-28; First posted 2016-05-19 (Estimated); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck; Locally Advanced; Squamous Cell Carcinoma; SCCHN; Untreated; High Risk; Intermediate Risk; Radiation Therapy; Cisplatin
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — pembrolizumab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Experimental): Cisplatin, Radiation, and Pembrolizumab started 3 weeks after completion of cisplating and radiation.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Radiation: IMRT
- Arm 2 (Experimental): Cisplatin and Radiation and Pembrolizumab given 1 week prior to the start of cisp/radiation and given every 3 weeks
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Radiation: IMRT

INTERVENTIONS:
Drug: Pembrolizumab — In both arms, the dose of pembrolizumab will be 200 mg (fixed dose) intravenous (IV) every 3 weeks for a total of 8 doses. In Arm 1, pembrolizumab will begin in week 10 of treatment, after cisplatin-IMRT is complete. In Arm 2, pembrolizumab will begin the week before cisplatin-IMRT.
  Other Names: Keytruda
Drug: Cisplatin — Patients will receive cisplatin once weekly as an IV infusion over 60 minutes, for a total of 7 doses, at the same time as radiation.
  Other Names: Platinol
Radiation: IMRT — IMRT will be delivered in 35 fractions (treatments) over 7 weeks (five treatments per non-holiday week) in one plan.

SUMMARY:
The goal of this research study is to learn which therapy order (adding pembrolizumab during vs. after cisplatin and radiation) may be more effective in treating head and neck cancer, as well as learn the side effects of these combinations. Pembrolizumab is an immune therapy, a drug that stimulates the immune system to fight cancer, and is FDA approved in lung cancer and melanoma.

DETAILED DESCRIPTION:
The study regimen consists of cisplatin and radiation for all patients, the standard treatment for head and neck cancer. All patients will also receive pembrolizumab (the study drug), and will be randomized to two treatment schedules: either pembrolizumab with cisplatin-radiation, or pembrolizumab after completing cisplatin-radiation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* If a woman of childbearing potential, documentation of negative pregnancy
* Histologically-confirmed head and neck squamous cell carcinoma with no evidence of distant metastasis. The primary site may be the oral cavity, oropharynx, larynx, or hypopharynx. Patients with squamous cell carcinoma of unknown primary, metastatic to cervical lymph nodes, are permitted to enroll.
* High risk or intermediate risk disease, defined below. Staging evaluation should be determined by imaging studies and complete head and neck exam in accordance with the American Joint committee on Cancer Staging Manual, 7th edition.

  o High risk patient must meet one of the following criteria:
* Surgically unresectable oral cavity. Patients who are technically resectable but refuse surgery due to morbidity (eg. total glossectomy) are also eligible. Medically inoperable patients are not eligible.
* Larynx: T4 any N; T2-3 and ≥ N2a
* Hypopharynx: T1-2N1-3 or T3-4N0-3
* Oropharynx: p16(-) AND T3-4 or ≥ N2a
* Unknown primary: p16(-) AND ≥ N2a

  o Intermediate risk patients must meet one of the following criteria:
* Oropharynx: p16(+) AND one of the following
* T3 or ≥ N2a AND ≥ 10 pack-years tobacco exposure (see Tobacco Assessment Form, Appendix A)
* T4 or N3 disease irrespective of tobacco exposure
* Unknown primary: p16(+) AND one of the following
* ≥ N2a AND ≥ 10 pack-years tobacco exposure
* N3 disease irrespective of tobacco exposure
* Patients must be untreated with curative-intent surgery for current diagnosis of Stage III, IVa, or IVb disease. Diagnostic biopsy of primary tumor and/or nodal sites is permitted.

  * Diagnostic simple tonsillectomy is permitted, provided patient has RECIST-measurable nodal disease.
  * Patients with a second HNSCC primary tumor are eligible for this study, provided more than 2 years have elapsed since the first diagnosis of HNSCC, the original tumor was managed with surgery only (no adjuvant chemotherapy or radiotherapy), and has not recurred.
* Patients with simultaneous primaries or bilateral tumors are excluded, with the exception of patients with bilateral tonsil cancers or patients with T1-2, N0, M0 differentiated thyroid carcinoma (resected or management deferred), who are eligible.
* No prior systemic (chemotherapy or biologic/molecular targeted therapy) or radiation treatment for head and neck cancer.

  * Patients may have received chemotherapy or radiation for a previous, curatively treated non-HNSCC malignancy, provided at least 2 years have elapsed.
  * Patients must be untreated with radiation above the clavicles.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Age ≥ 18
* Patients must have measurable disease according to RECIST 1.1
* Patients must demonstrate adequate organ function as defined.
* Sexually active patients must agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug.

Exclusion Criteria:

* Nasopharyngeal primary site
* Current participation in or previous participation in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment.
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational agent.
* Distant metastatic disease including CNS or leptomeningeal metastases is not allowed.
* History of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Received prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* History of second malignancy within 2 years prior to Study Day 1 (except for excised and cured non-melanoma skin cancer, carcinoma in situ of breast or cervix, superficial bladder cancer, or T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection).
* Active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.
* Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Received a live vaccine within 30 days prior to the first dose of trial treatment.
* Received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Significant pulmonary disease, including pulmonary hypertension, interstitial lung disease, or active, non-infectious pneumonitis.
* History or current evidence of any other medical or psychiatric condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Peripheral neuropathy ≥ Grade 2
* Significant cardiovascular disease, including:

  * Cardiac failure New York Heart Association (NYHA) class III or IV.
  * Myocardial infarction, severe or unstable angina within 6 months prior to Study Day 1.
  * History of serious arrhythmia (i.e., ventricular tachycardia, or ventricular fibrillation).
  * Ventricular cardiac arrhythmias requiring anti-arrhythmic medications.
  * Known left ventricular ejection fraction (LVEF) ≤ 50%.
* Significant thrombotic or embolic events within 3 months prior to Study Day 1.
* Major surgery within 6 weeks prior to Study Day 1 (subjects must have completely recovered from any previous surgery prior to Study Day 1). Biopsy, diagnostic tonsillectomy, airway tumor debulking or excisional lymph node biopsy do not constitute major surgery.
* Active infection requiring antibiotics or antifungals within 7 days prior to first dose of study drug.
* Significant electrolyte imbalance prior to enrollment (note that patients may be supplemented to achieve acceptable electrolyte values):

  * Hypomagnesemia <1.2 mg/dL or 0.5 mmol/L.
  * Hypokalemia < 3.0 mmol/L.
* Women must not be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Zandberg, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zandberg DP, Vujanovic L, Clump DA, Isett BP, Wang H, Sica G, Bao R, Li H, Ohr J, Skinner HD, Seethala RR, Chiosea SI, Ferris RL, Bauman JE. Randomized Phase II Study of Concurrent Versus Sequential Pembrolizumab in Combination With Chemoradiation in Locally Advanced Head and Neck Cancer. J Clin Oncol. 2025 Aug 10;43(23):2572-2582. doi: 10.1200/JCO-24-01580. Epub 2025 May 27. PMID 40424564
- [Derived] Ferris RL, Moskovitz J, Kunning S, Ruffin AT, Reeder C, Ohr J, Gooding WE, Kim S, Karlovits BJ, Vignali DAA, Duvvuri U, Johnson JT, Petro D, Heron DE, Clump DA, Bruno TC, Bauman JE. Phase I Trial of Cetuximab, Radiotherapy, and Ipilimumab in Locally Advanced Head and Neck Cancer. Clin Cancer Res. 2022 Apr 1;28(7):1335-1344. doi: 10.1158/1078-0432.CCR-21-0426. PMID 35091445

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin + Radiation + Pembrolizumab - Concurrent: Cisplatin and Radiation and Pembrolizumab given 1 week prior to the start of cisplatin and radiation and given every 3 weeks.
  Pembrolizumab: In both arms, the dose of pembrolizumab will be 200 mg (fixed dose) intravenous (IV) every 3 weeks for a total of 8 doses. In Arm 1, pembrolizumab will begin in week 10 of treatment, after cisplatin-IMRT is complete. In Arm 2, pembrolizumab will begin the week before cisplatin-IMRT.
  Cisplatin: Patients will receive cisplatin once weekly as an IV infusion over 60 minutes, for a total of 7 doses, at the same time as radiation.
  IMRT: IMRT will be delivered in 35 fractions (treatments) over 7 weeks (five treatments per non-holiday week) in one plan.
- Cisplatin + Radiation + Pembrolizumab - Sequential: Cisplatin, Radiation, and Pembrolizumab started 3 weeks after completion of cisplatin and radiation.
  Pembrolizumab: In both arms, the dose of pembrolizumab will be 200 mg (fixed dose) intravenous (IV) every 3 weeks for a total of 8 doses. In Arm 1, pembrolizumab will begin in week 10 of treatment, after cisplatin-IMRT is complete. In Arm 2, pembrolizumab will begin the week before cisplatin-IMRT.
  Cisplatin: Patients will receive cisplatin once weekly as an IV infusion over 60 minutes, for a total of 7 doses, at the same time as radiation.
  IMRT: IMRT will be delivered in 35 fractions (treatments) over 7 weeks (five treatments per non-holiday week) in one plan.
Period: Overall Study
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Started | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cisplatin + Radiation + Pembrolizumab - Concurrent: Cisplatin and Radiation and Pembrolizumab given 1 week prior to the start of cisplatin and radiation and given every 3 weeks
  Pembrolizumab: In both arms, the dose of pembrolizumab will be 200 mg (fixed dose) intravenous (IV) every 3 weeks for a total of 8 doses. In Arm 1, pembrolizumab will begin in week 10 of treatment, after cisplatin-IMRT is complete. In Arm 2, pembrolizumab will begin the week before cisplatin-IMRT.
  Cisplatin: Patients will receive cisplatin once weekly as an IV infusion over 60 minutes, for a total of 7 doses, at the same time as radiation.
  IMRT: IMRT will be delivered in 35 fractions (treatments) over 7 weeks (five treatments per non-holiday week) in one plan.
- Total: Total of all reporting groups
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.79 (7.55) | 63.64 (6.85) | 63.7184 (7.17250)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 37 | 38 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 39 | 35 | 74
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
ECOG [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) performance status (Score 0 - 4):
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    ECOG = 0 | 36 | 31 | 67
    ECOG = 1 | 4 | 8 | 12
    ECOG = 2 | 1 | 0 | 1
Stage [Count of Participants; unit: Participants] — NATIONAL CANCER INSTITUTE STAGING
  Stage 0 = Abnormal cells are present but have not spread to nearby tissue. Also called carcinoma in situ, or CIS. CIS is not cancer, but it may become cancer.
  Stage I, Stage II, and Stage III = Cancer is present. NOTE - The higher the number, the larger the cancer tumor and the more it has spread into nearby tissues.
  Stage IV = The cancer has spread to distant parts of the body. Higher stages indicate greater disease burden.
  Participants
    Stage = 3 | 3 | 1 | 4
    Stage = 4 | 34 | 32 | 66
    Not Stage 3 or 4 | 4 | 6 | 10
T Stage [Count of Participants; unit: Participants] — NATIONAL CANCER INSTITUTE STAGING - The T refers to the size and extent of the main tumor. The main tumor is usually called the primary tumor. Primary tumor (T) TX: Main tumor cannot be measured. T0: Main tumor cannot be found. T1, T2, T3, T4: Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T Stage = 1 | 1 | 1 | 2
    T Stage = 2 | 11 | 7 | 18
    T Stage = 3 | 10 | 10 | 20
    T Stage = 4 | 16 | 20 | 36
    T Stage = Not Available | 3 | 1 | 4
N Stage [Count of Participants; unit: Participants] — NATIONAL CANCER INSTITUTE TNM Staging System Regional lymph nodes (N) The N refers to the number of nearby lymph nodes that have cancer.
  NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1, N2, N3: Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer. Higher numbers indicate greater disease burden.
  Participants
    N Stage = 0 | 3 | 2 | 5
    N Stage = 1 | 1 | 5 | 6
    N Stage = 2 | 28 | 29 | 57
    N Stage = 3 | 6 | 2 | 8
    N Stage = Not Available | 3 | 1 | 4
Histology [Count of Participants; unit: Participants] — Classification of tissues and cells under a microscope.
  Participants
    Not applicable | 1 | 0 | 1
    SQUAMOUS CELL CA KERATINIZING, NOS | 1 | 0 | 1
    SQUAMOUS CELL CA METASTATIC, NOS | 2 | 2 | 4
    SQUAMOUS CELL CARCINOMA, NOS | 37 | 37 | 74
Primary Site [Count of Participants; unit: Participants]
  Hypopharynx | 4 | 1 | 5
  Larynx | 10 | 8 | 18
  Oropharynx | 27 | 30 | 57
p16 for oropharynx [Count of Participants; unit: Participants] — Patient status for presence of Human papillomavirus (HPV) strain p16
  Participants
    Negative for p16 for oropharynx | 16 | 17 | 33
    Positive for p16 for oropharynx | 22 | 21 | 43
    Not Available | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at ≤12 Months
Description: Probability of participants (expressed as a percentage) without disease progression at less than or equal to12 after start of treatment: Complete Response (CR) + Partial Response (PR)/total number of patients assessed. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 12 months
Population: All patients that received treatment and were radiologically evaluable for response.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 71 | 83

2. Primary Outcome: Progression-free Survival at ≤ 36 Months
Description: Probability of participants (expressed as a percentage) without disease progression at less than or equal to 36 months after start of treatment: Complete Response (CR) + Partial Response (PR)/total number of patients assessed. Per RECIST v1.1, CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 36 months
Population: All patients that received treatment and were radiologically evaluable for response.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 57 | 75

3. Primary Outcome: Progression-free Survival at ≤ 48 Months
Description: Probability of participants (expressed as a percentage) without disease progression time from treatment initiation to disease progression or death from any cause or last follow up. Per RECIST v1.1: Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 48 months
Population: All patients that received treatment and were radiologically evaluable for response.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 49 | 67

4. Primary Outcome: Acute Toxicity / DLT Rate
Description: The number of patients who experience unacceptable toxicity during protocol treatment as measured by the NCI CTCAE version 4.0
Time Frame: Up to 6 months
Population: All treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
Participants | 3 | 0

5. Primary Outcome: 1-year Locoregional Failure Rate
Description: Percent probability of participants for which time to locoregional failure (TTLRF) (calculated from treatment initiation to locoregional failure, or censored at other failure, death, or the last follow up; death is not an event) is less than 1 year. Locoregional failure is disease recurrence in either the location or regional location of the original disease, as opposed to a distant site.
Time Frame: Up to 1 year
Population: All treated patients.
Measure: Number; unit: percent probability of participants
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percent probability of participants | 15 | 4

6. Primary Outcome: 3-year Locoregional Failure Rate
Description: Percent probability of participants for which time to locoregional failure (TTLRF) (calculated from treatment initiation to locoregional failure, or censored at other failure, death, or the last follow up; death is not an event) is less than 3 years. Locoregional failure is disease recurrence in either the location or regional location of the original disease, as opposed to a distant site.
Time Frame: Up to 3 years
Population: All treated patients.
Measure: Number; unit: percent probability of participants
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percent probability of participants | 26 | 4

7. Secondary Outcome: Progression-free Survival (PFS)
Description: Median number of months from treatment initiation to disease progression or death from any cause or last follow up. Per RECIST v1.1 Progressive Disease: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: Up to 48 months
Population: All patients that received treatment and were radiologically evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
months | 37.00 [16.00 to NA] — Not reached due to insufficient number of participants with event of progression | NA [46.00 to NA] — Median not reached due to insufficient number of participants with event of progression

8. Secondary Outcome: Overall Survival (OS)
Description: The length of time from start of study treatment that patients are still alive.
Time Frame: Up to 48 months
Population: All patients on study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
months | NA [NA to NA] — Median not reached due to insufficient number of participants with event of death | NA [53.00 to NA] — Median not reached due to insufficient number of participants with event of death

9. Secondary Outcome: Overall Survival (OS) at ≤ 12 Months
Description: Probability of patients (expressed as a percentage) still alive at less than or equal to 12 months after start of study.
Time Frame: Up to12 months
Population: All patients on study.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 82 | 95

10. Secondary Outcome: Overall Survival (OS) at ≤ 36 Months
Description: Probability of patients (expressed as a percentage) still alive at less than or equal to 36 months after start of study.
Time Frame: Up to 36 months
Population: All patients on study.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 71 | 88

11. Secondary Outcome: Overall Survival (OS) at ≤ 48 Months
Description: Probability of patients (expressed as a percentage) still alive at less than or equal to 48 months after start of study.
Time Frame: Up to 48 months
Population: All patients on study.
Measure: Number; unit: percentage of patients
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
Number analyzed (Participants) | 41 | 39
percentage of patients | 71 | 83

ADVERSE EVENTS:
Time Frame: Up to 48 months
Description: Common Terminology Criteria for Adverse Events CTCAE (4.0) Serious Adverse Events = Grade 3 or greater events Advertising Events = events less than Grade 3
Arm/Group | Cisplatin + Radiation + Pembrolizumab - Concurrent | Cisplatin + Radiation + Pembrolizumab - Sequential
All-Cause Mortality (participants affected / at risk) | 11/41 | 6/39
Serious Adverse Events (participants affected / at risk) | 21/41 | 10/39
Other Adverse Events (participants affected / at risk) | 38/41 | 38/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation + Pembrolizumab - Concurrent (N=41) | Cisplatin + Radiation + Pembrolizumab - Sequential (N=39)
Anemia (Blood and lymphatic system disorders) | 4 | 0
Blood and lymphatic system disorders - Other, specifythrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyHypertension (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 2 | 2
General disorders and administration site conditions - Other, specifyDizziness (General disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyBacteremia (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyLung Infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifySepsis (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifypenumonia (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifypneumonia (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory, thoracic and mediastinal disorders - Other, specifypneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specifyCellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures - Other, specifyGJ Tube revision (Surgical and medical procedures) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Radiation + Pembrolizumab - Concurrent (N=41) | Cisplatin + Radiation + Pembrolizumab - Sequential (N=39)
Anemia (Blood and lymphatic system disorders) | 32 | 34
Blood and lymphatic system disorders - Other, specifygranulomatous lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Blood and lymphatic system disorders - Other, specifyvenous thrombosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specifyBradycardia (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyCAD (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyCoronary artery calcifications (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyMild aortic insufficiency (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifyMurmur (Cardiac disorders) | 0 | 1
Cardiac disorders - Other, specifySVC (left) (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifychronic obstructive pulmonary disease (Cardiac disorders) | 1 | 0
Cardiac disorders - Other, specifycoronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve disease (Cardiac disorders) | 0 | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 5 | 6
Sinus tachycardia (Cardiac disorders) | 15 | 11
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Ear and labyrinth disorders - Other, specifyEar Pressure (Ear and labyrinth disorders) | 1 | 0
Ear and labyrinth disorders - Other, specifyHearing Loss (Ear and labyrinth disorders) | 1 | 0
Ear and labyrinth disorders - Other, specifyItching Ears (Ear and labyrinth disorders) | 1 | 0
Ear and labyrinth disorders - Other, specifyOtotoxicity (Ear and labyrinth disorders) | 1 | 0
Ear and labyrinth disorders - Other, specifyRight Otalgia (Ear and labyrinth disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 5 | 6
Hearing impaired (Ear and labyrinth disorders) | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 12 | 7
Vertigo (Ear and labyrinth disorders) | 1 | 0
Endocrine disorders - Other, specifyDiabetes (Endocrine disorders) | 0 | 1
Endocrine disorders - Other, specifyTSH increased (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 3 | 5
Hypothyroidism (Endocrine disorders) | 15 | 11
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Bloating (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 20 | 20
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 11 | 11
Dry mouth (Gastrointestinal disorders) | 24 | 25
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2
Dysphagia (Gastrointestinal disorders) | 20 | 28
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specifyDry Heaves (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specifyFracture Tooth (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specifyGagging (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specifyGum Soreness (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specifyOdyNphagia (Gastrointestinal disorders) | 3 | 2
Gastrointestinal disorders - Other, specifyOral cavity erythema (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specifyOropharvngeal Pain (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specifyPain - swallowing (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, specifyodyNphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specifypNumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 24 | 24
Nausea (Gastrointestinal disorders) | 24 | 30
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 9 | 12
Salivary duct inflammation (Gastrointestinal disorders) | 18 | 18
Tooth development disorder (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 12
(General disorders) | 0 | 1
Chills (General disorders) | 2 | 2
Edema face (General disorders) | 1 | 0
Edema limbs (General disorders) | 2 | 0
Facial pain (General disorders) | 2 | 1
Fatigue (General disorders) | 22 | 21
Fever (General disorders) | 5 | 2
Flu like symptoms (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyBenign prostatic hyperplasia (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyErythema of throat (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyExcess phlegm (General disorders) | 1 | 0
Intermittent ear pain left side jaw/oral (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specifyPain in right neck/oral (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specifyThroat pain with swallowing (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specifyallergies seasonal (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifyintermittent L thigh pain (General disorders) | 1 | 0
intermittent ear, jaw left side pain (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specifyneuropathic pain (General disorders) | 0 | 1
General disorders and administration site conditions - Other, specifyodyNphagia (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifythroat pain (General disorders) | 1 | 0
General disorders and administration site conditions - Other, specifytumor bleeding (General disorders) | 1 | 0
Localized edema (General disorders) | 0 | 1
Neck edema (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 5 | 8
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Immune system disorders - Other, specifydecreased lymphocytes (Immune system disorders) | 1 | 1
Immune system disorders - Other, specifyseasonal allergies (Immune system disorders) | 1 | 0
Bladder infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyIncreased LDH (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyOral Thrush (Infections and infestations) | 2 | 1
Infections and infestations - Other, specifyOral thrush (Infections and infestations) | 0 | 1
Infections and infestations - Other, specifyRash-forearm itching (Infections and infestations) | 1 | 0
Infections and infestations - Other, specifyShingles (Infections and infestations) | 1 | 2
Infections and infestations - Other, specifyThrush (Infections and infestations) | 10 | 8
Infections and infestations - Other, specifyaspiration pneumonia (Infections and infestations) | 0 | 1
Infections and infestations - Other, specifyinfusion related reaction (Infections and infestations) | 0 | 1
Infections and infestations - Other, specifythrush (Infections and infestations) | 2 | 6
Lung infection (Infections and infestations) | 1 | 1
Mucosal infection (Infections and infestations) | 2 | 2
Phlebitis infective (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 20 | 19
Fall (Injury, poisoning and procedural complications) | 2 | 0
Injury, poisoning and procedural complications - Other, specifyInfusion Reaction (Injury, poisoning and procedural complications) | 0 | 1
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 3
Alkaline phosphatase increased (Investigations) | 3 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 3
Blood bilirubin increased (Investigations) | 2 | 0
CD4 lymphocytes decreased (Investigations) | 2 | 1
Cholesterol high (Investigations) | 3 | 6
Creatinine increased (Investigations) | 5 | 2
Hemoglobin increased (Investigations) | 1 | 0
INR increased (Investigations) | 0 | 1
Investigations - Other, specify (Investigations) | 0 | 1
Investigations - Other, specifyANC Decrease (Investigations) | 1 | 0
Investigations - Other, specifyAlanine AmiNtransferase decreased (Investigations) | 0 | 1
Investigations - Other, specifyBPH destruction (Investigations) | 0 | 1
Investigations - Other, specifyBUN elevation (Investigations) | 0 | 1
Investigations - Other, specifyBUN increased (Investigations) | 1 | 0
Investigations - Other, specifyBlisters (Investigations) | 1 | 0
Investigations - Other, specifyCreatine Clearance Increased (Investigations) | 1 | 0
Investigations - Other, specifyElevated BUN (Investigations) | 0 | 1
Investigations - Other, specifyIncreased Thyroid Peroxidase Antibodies (Investigations) | 0 | 1
Investigations - Other, specifyLDH Increase (Investigations) | 0 | 1
Investigations - Other, specifyLDH increase (Investigations) | 1 | 1
Investigations - Other, specifyLDH increased (Investigations) | 0 | 1
Investigations - Other, specifyLow testosterone (Investigations) | 1 | 1
Investigations - Other, specifyLyme Disease (Investigations) | 1 | 0
Investigations - Other, specifyRadionecrosis - Mouth (Investigations) | 1 | 0
Investigations - Other, specifyTSH increase (Investigations) | 0 | 1
Investigations - Other, specifyThrush (Investigations) | 0 | 1
Investigations - Other, specifyThyroid Peroxodase Ab (Investigations) | 1 | 0
Investigations - Other, specifyVitamin D deficiency (Investigations) | 0 | 1
Investigations - Other, specifyelevated TSH (Investigations) | 0 | 1
Investigations - Other, specifyfacial infection (Investigations) | 1 | 0
Investigations - Other, specifyhyperhydrosis (Investigations) | 1 | 0
Investigations - Other, specifyhyperlipidemia (Investigations) | 1 | 0
Investigations - Other, specifyoral thrush (Investigations) | 0 | 1
Investigations - Other, specifyradionecrosis (Investigations) | 0 | 1
Investigations - Other, specifysoft tissue nuerosis (Investigations) | 0 | 1
Investigations - Other, specifythyroid peroxidase antibodies (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 31 | 33
Lymphocyte count increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 22 | 19
Platelet count decreased (Investigations) | 22 | 22
Weight loss (Investigations) | 33 | 33
White blood cell decreased (Investigations) | 30 | 28
Anorexia (Metabolism and nutrition disorders) | 7 | 12
Dehydration (Metabolism and nutrition disorders) | 11 | 10
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hypernatremia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 5 | 6
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypokalemia (Metabolism and nutrition disorders) | 12 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 21 | 15
Hyponatremia (Metabolism and nutrition disorders) | 31 | 29
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 0
Metabolism and nutrition disorders - Other, specifyCachexia (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specifyDiabetes Type II (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specifyHYPERLIPIDEMIA (Metabolism and nutrition disorders) | 1 | 0
Metabolism and nutrition disorders - Other, specifyHypercholesterolemia (Metabolism and nutrition disorders) | 0 | 1
Metabolism and nutrition disorders - Other, specifyhypercholesterolemia (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal and connective tissue disorder - Other, specifyBilateral Upper Limb Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyCervical spondylosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyHeavy feet/stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyIntermittent left thigh pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyJaw Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyOA (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyParesthesia (Hands/ R Leg) (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyRadiation Fibrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyRib pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyRight Leg Pain Sciatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyRight Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifyRight neck stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specifySpinal SteNsis (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specifyThroat Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 8
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 2 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specifyAdrenal AdeNma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphonia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 9 | 7
Dysarthria (Nervous system disorders) | 0 | 1
Dysesthesia (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 26 | 31
Dysphasia (Nervous system disorders) | 6 | 4
Headache (Nervous system disorders) | 8 | 4
Movements involuntary (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specifyAutoNmic Insufficiency (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specifyNeuropathic pain (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specifyOdyNphagia (Nervous system disorders) | 1 | 1
Nervous system disorders - Other, specifyPresyncope (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specifySPINAL STENSIS (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specifydysosmia (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specifynumb right ear (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 3 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 2
Tremor (Nervous system disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 7 | 4
Depression (Psychiatric disorders) | 5 | 2
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 3
Restlessness (Psychiatric disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 2
Urinary frequency (Renal and urinary disorders) | 0 | 3
Urinary retention (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Prostatic obstruction (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other, specifyBenign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Reproductive system and breast disorders - Other, specifyBenign prostatic hypertrophy (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyCOPD (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Respiratory, thoracic and mediastinal disorders - Other, specifyEmphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyThroat erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyUlceration oropharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifyUpper Respiratoty Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifylung Ndules (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specifysob with exertion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 7
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify65cm open area Rt neck (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyBruising periorbital (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyDermatitis of right lower extremity (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyErythema Throat (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyNeck wound (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specifyPuritic skin (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other, specifyTape Burn to abd area (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specifyrash (Skin and subcutaneous tissue disorders) | 0 | 1
Surgical and medical procedures - Other, specifyinfusion siite extravastion (Surgical and medical procedures) | 0 | 1
Surgical and medical procedures - Other, specifytracheostomy site bleeding (Surgical and medical procedures) | 0 | 1
Surgical and medical procedures - Other, specifytumor bleeding (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 14 | 13
Hypotension (Vascular disorders) | 11 | 7
Lymphedema (Vascular disorders) | 5 | 7
Phlebitis (Vascular disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Vascular disorders - Other, specifyCoronary artery disease (Vascular disorders) | 0 | 1
Vascular disorders - Other, specifyLeft Ventricle Hypertrophy (Vascular disorders) | 0 | 1
Vascular disorders - Other, specifyVascular access complication (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-22): https://cdn.clinicaltrials.gov/large-docs/85/NCT02777385/Prot_SAP_000.pdf